CLINICAL TRIAL: NCT06054451
Title: Clinical Diagnosis and Pathological Spectrum of Porto-sinusoidal Vascular Disease in India
Acronym: PSVD-India
Status: Recruiting | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, ASSOCIATE PROFESSOR, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: IEC-INT/2023/MD-1081
Record Dates: First submitted 2023-08-11; First posted 2023-09-26 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Portal Hypertension; Budd-Chiari Syndrome; Non-Cirrhotic Portal Hypertension; Porto-Sinusoidal Vascular Diseases; Sinusoidal Obstruction Syndrome; Veno Occlusive Disease, Hepatic; Non-Cirrhotic Portal Fibrosis
Keywords: Porto-sinusoidal vascular disease; Budd Chiari Syndrom; extrahepatic portal venous obstruction; Portal Hypertension; Non-Cirrhotic Portal Fibrosis
MeSH Terms: conditions — Hypertension, Portal; Budd-Chiari Syndrome; Idiopathic Noncirrhotic Portal Hypertension; Hepatic Veno-Occlusive Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is a need to re-evaluate the patients classified as NCPH and determine whether the new histological classification proposed by the VALDIG applies to the Indian scenario. We intend to identify the patient cohorts who have been diagnosed as NCPH, NCPF, EHPVO, hepatic venous outlet tract obstruction (HVOTO), Veno-occlusive disease (VOD) and sinusoidal obstruction syndrome (SOS) based on their liver biopsy, endoscopy, HVPG, and radiology reports. These patients will be screened to find the patients who fit the diagnosis of PSVD. It is important to establish whether the new definition of PSVD is relevant to the Indian population and establish the usefulness of invasive tests like liver biopsy in diagnosing the disease. The patient cohorts meeting diagnosis of INCPH will be compared with those meeting the new diagnosis of PSVD. The investigators will describe the clinical (demographic, clinical risk factors, socioeconomic status), etiological (associated conditions, coagulation disorders medication use, genetic risk factors), imaging (based on ultrasound Doppler imaging or cross- sectional imaging), endoscopic, fibrosis tests (using non-invasive tests), and the histopathology of the patients who fulfil the criteria of PSVD.

DETAILED DESCRIPTION:
Portal hypertension is clinically characterized by a portal venous pressure gradient between the inferior vena cava and the portal vein is more than 5 mm. Liver cirrhosis remains the leading cause of portal hypertension in the western world. However, there are conditions where portal hypertension can even occur without liver cirrhosis, referred to as Noncirrhotic portal hypertension (NCPH). The term NCPH has been derived from a variety of histopathological entities such as hepatoportal sclerosis, noncirrhotic portal fibrosis, nodular regenerative hyperplasia, or incomplete septal fibrosis. In the absence of other causes of cirrhosis and portal venous thrombosis, the condition is termed idiopathic noncirrhotic portal hypertension. The histopathological findings of INCPH are not entirely specific to portal hypertension, similar changes can be seen in patients without portal hypertension. Therefore the term Porto-sinusoidal vascular disorder(PSVD) has been recently introduced to define a group of liver vessel disorders affecting the portal venules and sinusoids irrespective of the absence or presence of liver cirrhosis. This disease entity can have a varied clinical presentation and histological findings and has been associated with several immunological and systemic disorders.

Porto-sinusoidal vascular disease - Currently, for clinical practice, the VALDIG group has given a working definition for PSVD.

"Liver biopsy ≥20mm without cirrhosis with either 1 specific sign of portal hypertension OR 1 specific histological finding for PSVD" OR "Liver biopsy ≥20mm without cirrhosis with 1 sign not specific for portal hypertension AND 1 sign not specific for PSVD"

ELIGIBILITY:
Inclusion Criteria:

* Patients of 12-70 years, either gender with clinical, pathological radiological diagnosis of NCPH

Exclusion Criteria:

* Any patients having Cirrhosis based on clinical, pathological, or radiological diagnosis
* Any patients having active malignancy

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed as NCPF, EHPVO, HVOTO, SOS, VOD will be screened for reclassification based on diagnostic criteria for PSVD
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
To describe the clinical presentation of patients with a diagnosis of PSVD. | Day 0
  Listing clinical presentation (signs and symptoms) of patients with PSVD (variceal bleeding, pain, ascites, sensation of lump, etc)

SECONDARY OUTCOMES:
Radiological description of patients with PSVD based on CT venography | Day 0
  Radiological assessment will be done at baseline for characterization of changes of portal vein, small hepatic veins, liver and splenic morphology. Doppler of the portal vessels.
Radiological description of patients with PSVD based on Doppler Ultrasound | Day 0
  Radiological assessment will be done at baseline for characterization of changes of portal vein, small hepatic veins, liver and splenic morphology. Doppler of the portal vessels.
Histopathological features and subtypes of the PSVD spectrum in patients from India with assessment of parenchyma, vessels, portal triad and fibrosis | Day 0
  To classify the PSVD based on the histological finding the disease.
Ratio of liver stiffness and splenic stiffness using transient elastography in diagnosis of PSVD | Day 0
  To look for the trend of non-invasive techniques in PSVD such as ARFI, transient elastography, coagulation parameters, and inflammatory biomarkers in patients of PSVD
Change in biomarkers like Factor VIII Ag or vWF in diagnosis of PSVD | Day 0
  To look for the trend of non-invasive techniques in PSVD such as coagulation parameters, and inflammatory biomarkers in patients of PSVD
Presence of varices and other endoscopic findings in patients with PSVD | Day 0
  To look for esophageal varices and portal hypertensive gastropathy

CONTACTS AND LOCATIONS:
Overall Officials: Dr Madhumita Premkumar, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Dr. Madhumita Premkumar, Sector-12, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No